CLINICAL TRIAL: NCT02464839
Title: Prevalence and Clinical Characteristics of the Fungal Nail and Feet Infection in Patients With Hallux Valgus
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: Fungalhallux
Record Dates: First submitted 2015-04-30; First posted 2015-06-08 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Acquired Hallux Valgus
Keywords: Fungal nails and feet infection; Onychomycosis; Hallux valgus
MeSH Terms: conditions — Hallux Valgus; Onychomycosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hallux valgus patients: All of participants will perform a potassium hydroxide (KOH) examination and fungal culture to prove a fungal nail and feet fungal infection

SUMMARY:
This study was designed to demonstrate the prevalence of onychomycosis in hallux valgus patients. Additionally, all the prevalence of tinea pedis, the pattern of clinical manifestations, risk factors and coexistence foot deformities with hallux valgus were observed and recorded.

DETAILED DESCRIPTION:
Hallux valgus is an abnormal deviation of the big toe away from the midline of the body or toward the other toes of the foot that is associated especially with the wearing of ill-fitting shoes-compare bunion. According to the previous studies, the association of nails and feet of disorder such as superficial fugal foot infection, abnormal nail shape and onychomycosis was reported. Nevertheless, nail disorders have been neglected for examination and treatment due to asymptomatic clinical manifestations and low effects in quality of life, even though it is the common dermatologic problem in general population.

Nail disorders that coincidentally happen with foot deformities can cause by either onychomycosis or nail trauma. Unfortunately, clinical presentation of them is similar. Nevertheless onychomycosis is the common superficial fungal infection in Thai population. So that the empirical systemic treatment of onychomycosis in older patients by systemic therapy such as azoles group and terbinafine according to the standard regimen maybe induce serious side effects. If onychomycosis is suspected, the abnormal nail should be taken to confirm the diagnosis will be required. Therefore, this study was designed to demonstrate the prevalence of onychomycosis in hallux valgus patients. Additionally, all the prevalence of tinea pedis, the pattern of clinical manifestations, risk factors and coexistence foot deformities with hallux valgus were observed and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants was 18 years old or above.
* Participants were diagnosed hallux valgus foot deformity by specialists of physical medicine and rehabilitation based on clinical presentation at Foot Clinic, Siriraj hospital
* Participants accept the aim of this project and sign the consent form by themselves.

Exclusion criteria:

* Participants have other nail disorders before participate the research.
* Participants have the history of fungal infection treatment with one-month by topical or systemic therapy.
* Participants have coincidental bacterial infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed hallux valgus foot deformity by specialists of physical medicine and rehabilitation based on clinical presentation at Foot Clinic, Siriraj hospital
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The number of onychomycosis cases in hallux valgus patients | 4 months
  To record the number of onychomycosis cases in hallux valgus patients from date of first patients documented progression until the date of end of study. The data was analysed as percentage.

SECONDARY OUTCOMES:
The severity of onychomycosis in hallux valgus patients by using SCIO (Scoring Clinical Index for Onychomycosis) score at baseline | 4 months
  Patients with hallux valgus condition in this study were evaluated the severity of onychomycosis by using SCIO (Scoring Clinical Index for Onychomycosis) score at baseline.
The number of coexisting of tinea pedis cases with onychomycosis in hallux valgus patients | 4 months
  To record the number of coexisting of tinea pedis cases in hallux valgus patients from date of first patients documented progression until the date of end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Charussri - Leeyaphan, MD., Principal Investigator — Department of Dermatology Faculty of Medicine, Siriraj Hospital Mahidol University
Locations (1):
- Department of Dermatology, Bangkoknoi, Bangkok, Thailand